CLINICAL TRIAL: NCT06103643
Title: Simulation-based Emergency Brex Birth Management Training Impact on Students'Self Confidence and Competence
Brief Title: Simulation Based Emergency Brex Birth Management Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Ph.D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-732
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Birth
MeSH Terms: interventions — Models, Biological

STUDY DESIGN:
Intervention Model Description: parallel
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Reality Simulator (Experimental): Breech birth management training will be given by the responsible investigator, and then one of the groups will be allocated by randomization. Using High Reality Simulator will perform emergency breech birth. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.
  Interventions: Other: Using High Reality Simulator
- control group (Sham Comparator): Using model will perform emergency breech birth. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.
  Interventions: Other: Using High Reality Simulator

INTERVENTIONS:
Other: Using High Reality Simulator — Using High Reality Simulator will perform emergency breech birth.
  Other Names: model

SUMMARY:
The aim of this study is to determine the effect of SIMULATION-BASED EMERGENCY BREX BIRTH MANAGEMENT TRAINING IMPACT ON STUDENTS' SELF-CONFIDENCE AND COMPETENCE.

DETAILED DESCRIPTION:
Hypotheses H01; There was no difference between the students'self-confidence and competence of the simulation-based emergency brex birth management training group and students'self-confidence and competence score control group.

The study will be carried out in two different groups. The practice will start with meeting the students who apply to the study. After the students are evaluated in terms of eligibility criteria for the research, the students who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Breech birth management training will be given by the responsible investigator, and then one of the groups separated by randomization will perform emergency breech birth on the second group model using High Reality Simulator. These trainings will first be in the form of the instructor responsible for the groups demonstrating the application, and then the students will apply it one by one.

ELIGIBILITY:
Inclusion Criteria:

- Agreeing to participate in the research and obtaining written permission,

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Self-Confidence/Efficacy Scale in Patient Intervention | immediately before simulation and immediately after the training 2 months later
  It was developed by Jekins in America in 1983 for nursing students. The scale is used to describe students' perceptions of clinical decision-making based on their own statements (Jenkins, 2001).It was adapted into Turkish by Durmaz-Edeer and Sarıkaya (2015). The sub-dimensions of the scale, which consists of 40 items and four sub-dimensions; "Exploring options and ideas", "Inquiring into goals and values", "Evaluating consequences", and "Searching for information and impartially adopting new information". Each subscale consists of 10 items. The total score of the scale is between 40 and 200, and each subscale is scored between 10 and 50. There is no cutoff point on the scale. A high score from the scale indicates that the perception of decision-making is high, and a low score indicates that the perception of decision-making is low.The scale is evaluated based on each subscale and scale total score (Jenkins, 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye BAL, Study Director — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)